CLINICAL TRIAL: NCT03806010
Title: A Prospective Open Labelled Study to Evaluate if Central Sensitization as Measured With QST Alters Following Chronic Pain Interventions
Brief Title: QST and Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 15/LO/2094
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pain
Keywords: Quantitative sensory testing
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quantitative sensory testing: QST will be performed at baseline two weeks and 2 months
  Interventions: Procedure: Quantitative sensory testing

INTERVENTIONS:
Procedure: Quantitative sensory testing — Quantitative sensory testing

SUMMARY:
To establish the sensory profile of patients using quantitative sensory testing (QST) and questionnaires as well as the level of sensitisation using temporal summation and diffuse noxious inhibitory control paradigms in all patients undergoing a chronic pain intervention at Barts Health NHS Trust.

Primary objective- To identify the phenotype of responders and non-responders to a chronic pain intervention using QST sensory profile as well as the sensitisation paradigms.

Secondary objective- To establish the correlation between sensory profile, and sensitisation parameters as well as other measures of chronic pain as per Initiative on Methods, Measurement and Pain Assessment in clinical trials (IMMPACT) recommendation.

Common interventions performed at Barts Health NHS Trust includes Neuromodulation, targeted epidural steroid and/or radiofrequency treatment, 8% Capsaicin patch and pharmacological interventions such as anti-neuropathic agent and opioids.

ELIGIBILITY:
Inclusion Criteria:• Male and female patients between the age of 18-80 years who have a lumbar radiculopathy who have not undergone any spinal surgery.

* Minimum baseline pain rating of 50mm on a 100mm NRS in the painful area
* Chronic pain of at least 6 months
* Subject satisfies standard criteria in the study centre for SCS implantation and the NICE 159 criteria for management of intractable neuropathic pain.
* Subject satisfies standard criteria in the study centre for ONS implantation and the NICE 452 criteria for intractable chronic migraine.
* Patients who have given their written informed consent.
* Patient is able and willing to comply with study procedures and follow up schedule.

Exclusion Criteria:• Any inclusion criteria not met

* Female patients of childbearing age who is or plans on becoming pregnant during the course of the study
* Patients who have undergone radiofrequency or injection therapy at or on a target neural structure (DRG) during the past 90 days
* Patients with diabetes or any underlying neurological condition.
* Patients known to have a condition that in the investigator's judgment precludes participation in the study.
* Patients who have received an investigational drug or have used an investigational device in the 30 days preceding to study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain of at leasr 6 months
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
• To identify the phenotype of responders and non-responders to a chronic pain intervention using QST sensory profile as well as the sensitisation paradigms. | QST changes at 4 weeks is taken as primary objective.
  This is assessed by comparing and reporting any change in QST results before and after the intervention.

SECONDARY OUTCOMES:
• To establish the correlation between sensory profile and sensitisation parameters as well as other measures of chronic pain as per Initiative on Methods, Measurement and Pain Assessment in clinical trials (IMMPACT) recommendation • | 2 weeks 3, 6 months and one year
  QST changes
The effect on functionality and quality of life following chronic pain intervention | 2 weeks and 3, 6 months and 1 year.
  QST changes
Whether central sensitisation can be used as a bedside biomarker to predict outcome after interventions for chronic pain (i.e. the more centrally sensitised the more superior improvement from treatment) | 2 weeks and 3, 6 months and 1 year
  QST changes

CONTACTS AND LOCATIONS:
Overall Officials: vIVEK mEHTA, MD, Principal Investigator — Barts NHS Trust
Locations (1):
- Dr Theresa Wodehouse, London, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided